CLINICAL TRIAL: NCT03333226
Title: Axillary Reverse Mapping (ARM). Identification of the Arm Lymphatic Pathways in Breast Cancer Surgery to Prevent Breast Cancer Related Lymphedema (BCRL): a Randomized Clinical Trial.
Brief Title: Axillary Reverse Mapping (ARM) in Breast Cancer Surgery to Prevent Lymphedema. (ARMtrial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Paolo Carcoforo, MD, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RF-2013-02358165
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer Lymphedema
Keywords: Breast Neoplasms; Sentinel Lymph Node Biopsy; Lymph Node Excision; Technetium Tc 99m; Indocyanine Green; Lymphatic System; Secondary Prevention
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible patients for radioguided sentinel lymph node biopsy (rSLNB) will be randomly divided in two groups:
  1. experimental group in which all patients will be sent to both rSLNB and photodynamic Axillary Reverse Mapping (ARM) to evaluate the crossover between SLN and ARM lymph node. In case of SLN metastases, an ALND with ARM lymph node preservation will be performed.
  2. control group in which all patients will be sent to both rSLNB and photodynamic Axillary Reverse Mapping (ARM) to evaluate the crossover between SLN and ARM lymph node. In case of SLN metastases, an ALND with ARM lymph node removal will be performed.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be randomized before the SLNB procedure. Due to the type of intervention, the blinding of the treating surgeon will not be possible, thus the surgeon will be aware of both the intraoperative crossover between ARM lymph node and SLN (secondary outcome) and the allocation to ARM lymph node preservation or removal. Data about BCRL (primary outcome) will be collected by the physiatrist and the physiotherapist that will be blinded about the allocation (ARM lymph node preservation/removal) and the crossover between SLN of the breast and the arm's lymph node. The assessment of lymphoscintigraphic subclinical modification in the arm lymphatic drainage after SLNB and ALND (secondary outcomes) will be performed by a blinded nuclear medicine physician that will not be aware of the allocation (ARM lymph node preservation/removal) and the crossover between ARM lymph node and breast's SLN.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM lymph node preservation (Experimental): All patients will be sent to both rSLNB and photodynamic Axillary Reverse Mapping (ARM) to evaluate the crossover between SLN and ARM lymph node. In case of SLN metastases, an ALND with ARM lymph node preservation will be performed.
  Interventions: Procedure: Axillary Reverse Mapping (ARM)
- ARM lymph node removal (Active Comparator): All patients will be sent to both rSLNB and photodynamic Axillary Reverse Mapping (ARM) to evaluate the crossover between SLN and ARM lymph node. In case of SLN metastases, an ALND with ARM lymph node removal will be performed.
  Interventions: Procedure: Axillary Reverse Mapping (ARM)

INTERVENTIONS:
Procedure: Axillary Reverse Mapping (ARM) — ARM lymph node preservation versus removal

SUMMARY:
Breast cancer related lymphedema (BCRL) is a debilitating and distressing condition affecting approximately one out of five breast cancer survivors. BCRL is a chronic swelling of the upper arm following axillary lymph nodes dissection, and it is associated to a significant functional, psychological and social morbidity, with an heavy impact on life quality. Several studies reported BCRL incidence between 6.7% and 62.5% for different population cohorts. Randomized clinical trials (RCTs) reported that sentinel lymph node biopsy (SLNB) when compared with axillary lymph node dissection (ALND) leads to a significant reduction in postoperative complications. However, the advent of SLNB does not solve the problem of BCRL with a concrete chance to develop a lymphedema after single SLNB around 7%. Health care cost of BCRL rehabilitative treatment is not available in literature yet. Few studies considered incidence, risk factors and treatment costs of BCRL among working-age women after breast cancer treatment, reporting that BCRL population had significantly higher rehabilitative medical costs ($14,877 to $23,167) with twice as much risk to develop BCRL complications, such as lymphangitis or cellulitis when compared to "BCRL free" population (OR = 2.02, P = .009).

Axillary reverse mapping (ARM) procedure claims to map and preserve arm lymphatic drainage during ALND and/or during SLNB, reducing BCRL development. ARM is developed as result of assumption that arm's lymphatic pathway is not involved by metastatic tumor cells of the primary breast cancer. However, when the arm lymph node correspond to the SLN it should be removed for correct tumor staging, thus a lymphatic drainage disruption onset will be expected with BCRL risk increase.

During the ARM procedure, a fluorescence imaging technique (photodynamic procedure) is useful for detecting lymphatic drainage of the upper limb and it allows in differentiating the fluorescent ARM node from the SLN identified by the radioguided technique (99mTC-Nanocoll).

DETAILED DESCRIPTION:
The investigators will conduct a randomized clinical trial (RCT) at the S. Anna University Hospital of Ferrara (Italy) on consecutive patients undergoing SLNB for breast cancer and subsequent ALND in case of SLN metastases. Eligible patients for radioguided sentinel lymph node biopsy (rSLNB) will be randomly divided in two groups: 1) experimental group in which patients undergoing rSLNB and ARM photodynamic procedure; and, in case of SLN metastases, subsequent ALND with ARM node preservation; 2) control group in which patients undergoing rSLNB and ARM photodynamic procedure; and, in case of SLN metastases, subsequent ALND with ARM node removal.

Consent procedure

Patients will be visited in the outpatient clinic by one of the treating surgeon, who will approach the subject and explain the study. If the patient is interested in participating, further details will be provided and consent will be obtained.

Experimental design

Step 1

Patients enrolled in both groups will be subjected to rSLNB associated to ARM photodynamic procedure.

Radioguided SLNB technique:

The day before surgery, four peri-areolar subcutaneous injections of Tc-99m Nanocoll® will be performed for an overall volume of 0.4 ml (standard activity of 74 MBq). Pre-operative imaging of SLN consists of an anterior and lateral static acquisition, generally performed between 1 and 5 hours post-injection (max. 18 hours), by means of a double head gammacamera (Siemens, ECAM). The gamma camera energy selection peak is centered on the 140 KeV of 99mTc (with a window of ± 10%), and the use of high-resolution collimators and of a 256x256 acquisition matrix. Acquisition time varies between 2 and 8 minutes. Cutaneous projection of SLN will be marked with a skin-marking pen. The day of surgery, after intraoperative routine prep and drape, a handheld gamma probe (EuroProbe III, EURORAD, Chennevières-sur-Marne, France) will be used to localize radioactivity before skin incision and during axillary dissection to identify SLN, that is defined by counts >10% of background.

ARM photodynamic procedure:

The day of surgery, 15 minutes before surgical incision, patients will be subjected to injection of 1 ml of ICG (5mg/ml) in the upper forearm and during SLNB we will perform an evaluation of lymphatic arm pathways with fluorescence (IC-Flow Diagnostic Green, SEDA S.p.a., Milano, Italy). If a crossover between SLN of the breast and the arm's lymph node will be find, the ARM lymph node identified by the photodynamic technique will be excised for pathological evaluation.

Step 2

Patients with tumor positive SLN, eligible for ALND, will undergo to preoperative arm lymphoscintigraphy in order to asses possible changes in lymphatic drainage pathways of the arm after rSLNB.

The day before ALND, an injection of a volume of 0.4 ml of Tc-99m Nanocoll® in each hand will be performed, fractioned in all interdigital space. The subsequent scintigraphic planar acquisition is performed using a double head gamma-camera (Siemens, Ecam) according the following protocol:

* 5 minutes post injection: imaging acquisition on hands and forearms positioned over collimator with a marker near right arm;
* 10 minutes post injection :anterior acquisition with gamma camera head 1 on elbows and shoulders;
* 15 minutes post injection : anterior acquisition on both axilla and thorax using cobalt wires markers drawing cranium profile;
* 20 minutes post injection :marking with skin-marking pen of skin projection of most radioactive axillary nodes;
* 120/180 minutes post injection : acquisition in the same position for checking of possible number and/or site changes of nodes marked before.

Step 3

Experimental group:

In case of SLN metastases, during radical ALND (I, II,III levels of Berg), the ARM lymph node identified with both radioguided and photodynamic methods will be isolated from the other axillary lymph nodes and preserved. Photodynamic method will also allow us to visualize the lymphatic drainage of the arm that will be preserved.

Control group:

In case of SLN metastases, during radical ALND (I, II,III levels of Berg), the ARM lymph node identified with both radioguided and photodynamic method will be isolated from the other axillary lymph nodes and removed.

Step 4

The post-operative follow up will be conducted in inpatient setting and after discharge in outpatient setting (surveillance for early and delayed surgical complications). All patients will be clinically evaluated at 10, 30, 60, and 180 days after surgery and undergoing bilateral arms lymphoscintigraphy at 60 days after surgery to determine possible lymphoscintigraphic changes underlying a subclinical BCRL. Clinically follow-up will include the clinical presentation (pain, integumentary abnormalities, paresthesia, hypoesthesia, neuro-vascular deficits), measurement of 7 records [diameters of the upper limb (hand, wrist, 15 cm and 10 cm distally to olecranon, elbow (olecranon), 10 cm and 15 cm proximally to olecranon)] and final conversion into volumes. In case of BCRL diagnosis patients will be addressed to rehabilitative center for therapy.

Statistical analysis

A prospective analysis will be obtained from database in which patients data will be collected, with details of the patients and tumors characteristics, lymphatic drainage of the upper extremity, intra- and post-operative outcome, and follow up. The power analysis, based on preliminary results, reports that 150 women in each group are required to achieve a power of 0.9 and to detect a significant difference (p<0.05). Data will be expressed as mean ± standard deviation or median (interquartile range - IQR 25-75) according to the distribution. The Shapiro-Wilk test will be used to assess the assumption of normality. Categorical data will be presented as number (%). Data will be analyzed using the Chi-square test to compare percentages, t-Student test will be used to compare the means and Mann-Whitney test to compare non parametric data. Logistic regression analysis will be employed to construct a model predicting BCRL using factors regarding the patient [age, gender, BMI, American Society of Anesthesiology (ASA) classification], the tumor (size, stage, bio-molecular characteristics ), crossover, type of intervention (preservation of ARM lymph node vs. dissection), and post-operative treatment (chemotherapy, radiotherapy). Significance will be considered for values of p<0.05. Statistical analysis will be performed with IBM SPSS Statistics for Windows, Version 24.0 (IBM Corp. Armonk, NY: IBM Corp.).

ELIGIBILITY:
Inclusion Criteria:

* T1-T2 stage breast cancer

Exclusion Criteria:

* axillary lymph node metastasis;
* previous surgery on the ipsilateral axilla;
* neoadjuvant chemo-radiotherapy;
* presence of primitive lymphedema of the arm;
* allergy to Iodine, thyroid disease, renal and hepatic impairment (for issues related to Indocyanine Green)
* pregnancy;
* patients refusing to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Breast Cancer Related Lymphedema (BCRL) after Axillary Lymph Node Dissection (ALND) | From the day of surgery to 12 months after surgery
  Incidence of BCRL in patients in whom the ARM lymph node is preserved compared to those in which it is removed. Clinically follow-up will include the clinical presentation (pain, integumentary abnormalities, paresthesia, hypoesthesia, neuro-vascular deficits), standardized measurement of 7 records [diameters of the upper limb (hand, wrist, 15 cm and 10 cm distally to olecranon, elbow (olecranon), 10 cm and 15 cm proximally to olecranon)] and final conversion into volumes.

SECONDARY OUTCOMES:
Incidence of Breast Cancer Related Lymphedema (BCRL) after Sentinel Lymph Node Biopsy (SLNB) alone | From the day of surgery to 12 months after surgery
  Clinically follow-up will include the clinical presentation (pain, integumentary abnormalities, paresthesia, hypoesthesia, neuro-vascular deficits), standardized measurement of 7 records [diameters of the upper limb (hand, wrist, 15 cm and 10 cm distally to olecranon, elbow (olecranon), 10 cm and 15 cm proximally to olecranon)] and final conversion into volumes.
Crossover between Sentinel Lymph Node (SLN) of the Breast and the ARM lymph node | Intraoperatively
  Intraoperatively, the radioguided technique (Tc-99m Nanocoll) will be used to identify the SLN of the breast; at the same time, the Axillary Reverse Mapping (ARM) of the upper limb will be carried out by Indocyanine Green, and the ARM lymph node will be identified and preserved. If a crossover between SLN of the breast and the arm's lymph node will be find, the ARM lymph node identified by the photodynamic technique will be excised for pathological evaluation.
Lymphoscintigraphic sub-clinical modifications of arm lymphatic drainage after ALND | The day before ALND and at 60 days after ALND
  Bilateral arms lymphoscintigraphy

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria S. Anna, Cona, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Formal requests will be evaluated.

REFERENCES:
- [Background] Sakorafas GH, Peros G, Cataliotti L, Vlastos G. Lymphedema following axillary lymph node dissection for breast cancer. Surg Oncol. 2006 Nov;15(3):153-65. doi: 10.1016/j.suronc.2006.11.003. Epub 2006 Dec 21. PMID 17187979
- [Background] McWayne J, Heiney SP. Psychologic and social sequelae of secondary lymphedema: a review. Cancer. 2005 Aug 1;104(3):457-66. doi: 10.1002/cncr.21195. PMID 15968692
- [Background] Purushotham AD, Upponi S, Klevesath MB, Bobrow L, Millar K, Myles JP, Duffy SW. Morbidity after sentinel lymph node biopsy in primary breast cancer: results from a randomized controlled trial. J Clin Oncol. 2005 Jul 1;23(19):4312-21. doi: 10.1200/JCO.2005.03.228. PMID 15994144
- [Background] Wilke LG, McCall LM, Posther KE, Whitworth PW, Reintgen DS, Leitch AM, Gabram SG, Lucci A, Cox CE, Hunt KK, Herndon JE 2nd, Giuliano AE. Surgical complications associated with sentinel lymph node biopsy: results from a prospective international cooperative group trial. Ann Surg Oncol. 2006 Apr;13(4):491-500. doi: 10.1245/ASO.2006.05.013. Epub 2006 Mar 2. PMID 16514477
- [Background] Shih YC, Xu Y, Cormier JN, Giordano S, Ridner SH, Buchholz TA, Perkins GH, Elting LS. Incidence, treatment costs, and complications of lymphedema after breast cancer among women of working age: a 2-year follow-up study. J Clin Oncol. 2009 Apr 20;27(12):2007-14. doi: 10.1200/JCO.2008.18.3517. Epub 2009 Mar 16. PMID 19289624
- [Background] Ponzone R, Mininanni P, Cassina E, Sismondi P. Axillary reverse mapping in breast cancer: can we spare what we find? Ann Surg Oncol. 2008 Jan;15(1):390-1; author reply 392-3. doi: 10.1245/s10434-007-9663-6. Epub 2007 Nov 8. No abstract available. PMID 17990039
- [Background] Boneti C, Korourian S, Diaz Z, Santiago C, Mumford S, Adkins L, Klimberg VS. Scientific Impact Award: Axillary reverse mapping (ARM) to identify and protect lymphatics draining the arm during axillary lymphadenectomy. Am J Surg. 2009 Oct;198(4):482-7. doi: 10.1016/j.amjsurg.2009.06.008. PMID 19800452
- [Background] Britton TB, Solanki CK, Pinder SE, Mortimer PS, Peters AM, Purushotham AD. Lymphatic drainage pathways of the breast and the upper limb. Nucl Med Commun. 2009 Jun;30(6):427-30. doi: 10.1097/MNM.0b013e328315a6c6. PMID 19319006
- [Background] Noguchi M, Noguchi M, Nakano Y, Ohno Y, Kosaka T. Axillary reverse mapping using a fluorescence imaging system in breast cancer. J Surg Oncol. 2012 Mar;105(3):229-34. doi: 10.1002/jso.22094. Epub 2011 Sep 12. PMID 21913193
- [Background] Han C, Yang B, Zuo WS, Zheng G, Yang L, Zheng MZ. The Feasibility and Oncological Safety of Axillary Reverse Mapping in Patients with Breast Cancer: A Systematic Review and Meta-Analysis of Prospective Studies. PLoS One. 2016 Feb 26;11(2):e0150285. doi: 10.1371/journal.pone.0150285. eCollection 2016. PMID 26919589
- [Background] Yue T, Zhuang D, Zhou P, Zheng L, Fan Z, Zhu J, Hou L, Yu F, Dong X, Xiao L, He Q. A Prospective Study to Assess the Feasibility of Axillary Reverse Mapping and Evaluate Its Effect on Preventing Lymphedema in Breast Cancer Patients. Clin Breast Cancer. 2015 Aug;15(4):301-6. doi: 10.1016/j.clbc.2015.01.010. Epub 2015 Feb 19. PMID 25776198
- [Background] Sarri AJ, Dias R, Laurienzo CE, Goncalves MC, Dias DS, Moriguchi SM. Arm lymphoscintigraphy after axillary lymph node dissection or sentinel lymph node biopsy in breast cancer. Onco Targets Ther. 2017 Mar 6;10:1451-1457. doi: 10.2147/OTT.S117830. eCollection 2017. PMID 28331338